CLINICAL TRIAL: NCT05456269
Title: An Open-label Two Strata Study of Bisantrene in Combination With Cytarabine Arabinoside or Bisantrene in Combination With Oral Decitabine/Cedazuridine for the Treatment of Acute Myeloid Leukemia Patients With Extramedullary Disease
Brief Title: A Study of Bisantrene Combined With Cytarabine or With Decitabine for Adult Subjects With Extramedullary AML and MDS
Acronym: BISECT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: commercial reason
Sponsor: Race Oncology Ltd (Industry)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RAC-006
Record Dates: First submitted 2022-07-04; First posted 2022-07-13 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Higher Risk Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
Keywords: combination treatment intervention
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — bisantrene; Cytarabine; Arabinofuranosylcytosine Triphosphate; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratum 1 (Experimental): Bisantrene infused daily for 7 days of induction cycle 1; followed by bisantrene infusion on Days 1 and 2 and cytarabine arabinoside continuous infusion on Days 1 to 5 of each consolidation cycle for up to 3 cycles.
  Each cycle is 28 days, with a potential to expand to 42 days to allow for full hematologic recovery.
  Interventions: Drug: Bisantrene Dihydrochloride (high dose); Drug: Cytarabine Hydrochloride
- Stratum 2 (Experimental): Decitabine/cedazuridine daily on Days 1-5, Bisantrene infusion on Days 3 and 5 in 28 day cycle. Treatment repeats every 28 days up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Each has potential to expand to 42 days to allow for full hematologic recovery.
  Interventions: Drug: Bisantrene Dihydrochloride (low dose); Drug: Decitabine and cedazuridine

INTERVENTIONS:
Drug: Bisantrene Dihydrochloride (high dose) — Induction monotherapy cycle: IV bisantrene daily on Days 1 to 7, starting at 250 mg/m2 then adjusted to either 275 mg/m2 or 225 mg/m2 based on confirmed dose (Run-in) Consolidation combination cycle/s: IV bisantrene daily on Days 1 to 2
  Other Names: RC110; Zantrene®; Xantrene®
  Arms: Stratum 1
Drug: Bisantrene Dihydrochloride (low dose) — IV bisantrene at escalating doses for 3 dose levels of 50, 65, 85 mg/m2 on Days 3 and 5 until Maximum tolerated dose (MTD) reached.
  Other Names: RC110; Zantrene®; Xantrene®
  Arms: Stratum 2
Drug: Cytarabine Hydrochloride — Consolidation cycles: continuous IV cytarabine (100mg/m2) on Days 1 to 5
  Other Names: Ara-C; Cytarabine arabinoside; Cytosar-U®
  Arms: Stratum 1
Drug: Decitabine and cedazuridine — PO fixed-dose decitabine/cedazuridine 35/100 mg tablet daily for 5 days (Days 1 to 5), 1 hour prior bisantrene infusion
  Other Names: ASTX727
  Arms: Stratum 2

SUMMARY:
This is a two strata Phase 1b study to assess the safety and efficacy of bisantrene (RC110) in combination with a) cytarabine arabinoside (Ara-C) treatment for patients with relapsed or refractory (R/R) Acute Myeloid Leukemia (AML) with extramedullary disease and able to tolerate intensive chemotherapy; b) in combination with decitabine/cedazuridune (ASTX727) new or relapsed or refractory AML or high risk MDS or CMML with extramedullary disease and unable or not willing to have intensive chemotherapy.

DETAILED DESCRIPTION:
The study is a multicenter, open label in patients with haematological malignancy / myeloproliferative disease (AML, MDS and CMML) and extramedullary disease (EMD) investigating 2 treatment regimens:

1. Stratum 1 will investigate use of high dose intravenous (IV) bisantrene (RC110) in combination with IV Ara-C for R/R AML with EMD able to tolerate intensive chemotherapy. This includes a run-in stage to confirm the dose of bisantrene (RC110) for induction and in combination with Ara-C for consolidation cycles and an expansion and an expansion stage that will treat additional patients at the confirmed bisantrene dose for induction and in combination with Ara-C consolidation cycles;
2. Stratum 2 will investigate use lower doses intravenous (IV) bisantrene (RC-110) in combination with fixed-dose oral decitabine/cedazuridine (ASTX727) to determine the maximum tolerated dose (MTD) for new or R/R AML and HR-MDS/CMML unable to tolerate intensive chemotherapy.

Pre-screening will be conducted to identify patients with EMD diagnosed by standard clinical practice including histology and by fluorine-18-fluorodeoxyglucose positron emission tomography/computed tomography (18F FDG-PET/CT) imaging.

ELIGIBILITY:
Inclusion Criteria:

[Both Stratums]

1. Patients must be able to understand and provide informed written consent.
2. Patients must be of age ≥ 18 years at the time of signing the informed consent.
3. Extramedullary disease (i.e., AML) by 18F-FDG PET/CT and/or clinical morphology (histopathology of chloroma, leukemia cutis or AML) at pre-screening
4. Patients who have undergone stem cell transplantation (SCT), maybe included if they are ≥ 8 weeks from stem cell infusion (autologous or allogeneic), have no active graft versus host disease (GVHD), are off immune suppression for at least 2 weeks, and do not have a history of veno occlusive disease (VOD).
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.0 for intensive Stratum 1 patients and ≤ 3.0 for low intensity treatment Stratum 2 patients.
6. Life expectancy estimated to be > 3 months.
7. Adequate organ function as evidenced by serum total bilirubin ≤ 2.0 mg/dL, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 × the upper limit of normal (ULN), serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance of ≥ 60 mL/min.
8. Cardiac ejection fraction ≥ 50%, assessed by 2-Dimensional (2D) echocardiogram.
9. Females of childbearing potential must have a negative serum pregnancy test at enrolment or within 14 days before study entry and must agree to use an adequate method of contraception, i.e., barrier method, during the study until 30 days after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception, i.e., barrier method, during the study until 30 days after the last treatment.

   [Stratum 1 only]
10. Diagnosis of R/R AML, defined as ≥ 5% blasts in a patient with known prior history of AML according to World Health Organization (WHO) criteria. Patients with AML that have relapsed at least once or are primary induction failure will be eligible.

    [Stratum 2 only]
11. Patients with diagnosis of de novo AML with EMD, or R/R AML with EMD.
12. Patients with MDS or CMML, diagnosed according to the 2016 WHO classification with high-risk disease per the International Prognostic Scoring System (IPSS) of intermediate 2 or higher for both MDS and CMML. Revised IPSS intermediate risk patients can be considered after discussion with the Investigator.

Exclusion Criteria:

[Both Stratums]

1. Acute promyelocytic leukemia (APML) M3 subtype of AML.
2. Central nervous system manifestations of AML, unless treated and with no residual manifestations (either by cerebrospinal fluid (CSF) cytology, radiologically or by other clinical assessments) in the last 2 weeks.
3. Evidence or recent history of CNS disease, including primary or metastatic brain tumors, seizure disorders unless there is evidence for clearance of CNS leukemia (2 leukemia free CSFs by morphology and /or flow cytometry 1 week apart).
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cirrhosis, chronic obstructive or restrictive pulmonary disease, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
5. Other active malignancy (including other hematologic malignancies) or other malignancy within the last 12 months except non-melanoma skin cancer or cervical intraepithelial neoplasia.
6. Major surgery within 4 weeks of treatment.
7. Any medical, psychological, or social condition that may interfere with study patient or compliance or may compromise the patient's safety in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Stratum 1, Stage 1: Dose confirmation | 8 weeks
  Maximum tolerated dose (MTD) based on occurence dose limiting toxicity (DLT) graded according to the National Cancer Institute Common Terminology Criteria (NCI CTCAE) for Adverse Events v5.0 after completion of 2 cycles of treatment
Stratum 1 Stage 2: Overall response | 4 weeks
  Morphological overall response, defined as complete remission (CR), CR with incomplete hematologic recovery or morphologic leukemia free state (MLFS), after completion of first treatment cycle 1
Stratum 2: Safety and tolerabillity | 4 weeks
  Assessed based on the occurence of non-hematological Dose limiting toxicity (DLT) as graded according to the National Cancer Institute Common Terminology Criteria (NCI CTCAE) for Adverse Events v5.0 at the completion of cycle 1.

SECONDARY OUTCOMES:
Stratum 1: Minimal Residual Disease (MRD) response | 4 weeks
  Response is defined as MRD negativity with and without morphological complete remission (CR), at low level molcular MRD with CR and MRD relapse (coversion MRD negativity to positivity) at the completion of cycle 1
Stratum 1: Radiologic response | 4, 8 and 16 weeks
  Response evaluation by 18F-FDG-PET/CT is based on the 5-point scale Deauville criteria for complete metabolic response (defined as Deauville Score (DS) 1, 2, or 3) or for partial metabolic response (defined DS of 4 or 5 with decrease in number or activity in bone marrow/EMD disease at the completion of cycles 1,2 and 4..
Stratum 1: Dermal clinical response | 4, 8, 12, and 16 weeks
  Dermal response based on improvement on the static investigator global assessment (IGA) 5-point disease severity scores, where higher score indicate more disease, defined as decrease of at least two points relative to baseline at the completion of cycles 1,2 3 and 4.
Stratum 1: Dermal therapeutic response | 4, 8, 12, and 16 weeks
  Dermal therapeutic improvement based on the static investigator global assessment (IGA) 5-point disease severity scores, where higher score indicate more disease, defined as decrease of at least two points relative to baseline at the completion of cycles 1,2 3 and 4.
Stratum 1: Safety and tolerability | 4, 8, 12 and 16 weeks
  Safety and tolerability based on the incidence and severity of adverse events assessed using National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0, grade per event, patient, and cycle of treatment.
Stratum 1: Number of participants that recieve subsequent allogeneic hematopoietic stem cell transplant | 5 years
  Proportion of patients who receive subsequent allogeneic HSCT
Stratum 1:Event free survival (EFS) | Day 1 (treatment start) to 5 years
  EFS assessed between treatment start until the date of the earliest of these events: death, progression or off protocol-treatment for any reason using the Kaplan-Meier method
Stratum 1: Overall Survival (OS) | Day 1 (treatment start) to 5 years
  OS assessed between treatment start until death due to any cause using the Kaplan-Meier method
Stratum 2: Overall response | 4 weeks
  Morphological overall response, defined as either CR or CR as complete remission (CR), CR with incomplete hematologic recovery, CR with incomplete count recovery or MLFS. For patients with MDS/CMML, overall response, defined as either CR or modified CR mCR with haematological improvement (HI) at the end of cycle 1
Stratum 2: Minimal Residual Disease (MRD) response | 16 weeks
  Response is defined as MRD negativity with and without morphological complete remission (CR), at low level molecular MRD with CR and MRD relapse (coversion MRD negativity to positivity) at the completion of cycle 4.
Stratum 2: Radiologic response | 16, 36 and 48 weeks
  Response evaluation by 18F-FDG-PET/CT, based on the 5-point scale Deauville criteria for complete metabolic response (defined as as Deauville Score (DS) 1, 2, or 3) or for partial metabolic response (defined as DS of 4 or 5 with decrease in number or activity in bone marrow/EMD disease) at the the completion of cycles 4, 6, 9 and 12
Stratum 2: Dermal clinical response | 4, 24, 36 and 48 weeks
  Dermal clinical improvement based on the static investigator global assessment (IGA) 5-point disease severity scores, where higher score indicate more disease, defined as as disease severity score of 1 (almost clear) or 0 (clear) and at least a two grade/point decrease in severity score relative to baseline the completion of cycles 4, 6, 9 and 12
Stratum 2: Dermal therapeutic response | 4, 24, 36 and 48 weeks
  Dermal therapeutic improvement based on the static investigator global assessment (IGA) 5-point disease severity scores, where higher score indicate more disease, defined as decrease of at least two points relative to baseline the completion of cycles 4, 6, 9 and 12.
Stratum 2: Event free survival (EFS) | Day 1 (treatment start) up to 5 years
  EFS assessed between treatment start until the date of the earliest of these events: death, progression or off protocol-treatment for any reason assessed
Stratum 2: Overall survival (OS) | Day 1 (treatment start) to 5 years
  OS assessed between treatment start until death due to any cause using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Marinella Messina, PhD, Study Director — Clinical Director
Locations (1):
- Calvary Mater, Newcastle, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No